CLINICAL TRIAL: NCT03629535
Title: Accuracy of Non-invasive Non-oscillometric Blood Pressure Wristband
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 17-00884
Record Dates: First submitted 2018-08-09; First posted 2018-08-14 (Actual); Results first posted 2021-02-02 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2021-01

CONDITIONS: Hypotension; Hypertension
MeSH Terms: conditions — Hypotension; Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Patients in SICU (Experimental): Patients in the SICU with an intra-arterial blood pressure monitor already in place will be considered as subjects.
  Interventions: Device: Non-invasive non-oscillometric blood pressure wristband device; Device: Invasive intra-arterial blood pressure monitors.

INTERVENTIONS:
Device: Non-invasive non-oscillometric blood pressure wristband device — The device is a band intended to be worn on the wrist for intermittent blood pressure measurements. The device applies no inflatable mechanics or moving parts. The wristband is watertight and can be worn as any type of bracelet.
Device: Invasive intra-arterial blood pressure monitors. — Because the subjects also have an intra-arterial blood pressure monitor in place, the subjects will serve as their own control

SUMMARY:
The primary objective of the present investigation is to determine the accuracy of a non-invasive non-oscillometric blood pressure wristband device when compared to invasive intra-arterial blood pressure monitors. In an intensive care unit patients who already have an intra-arterial blood pressure monitor in place, this wristband device will be applied and blood pressure readings compared for approximately 15 minutes. Blood pressure readings will be gathered and compared.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to the Surgical Intensive Care Unit who are already fitted with an invasive Arterial Line (A- Line) are eligible for the trial, and no volunteers candidates for an A Line are requested.

Exclusion Criteria:

* Within the candidate group of individuals whose procedure in the hospital requires an A-Line, the wristband may not, for various reasons, produce a clean signal. This is immediately determined after wearing the band (and may be related to the size of the wrist of the subject, among other things). Such candidates will be excluded from admission to the study.
* All data from a subject shall be excluded if the invasive reference systolic blood range is greater than 20 mmHg (2, 67 kPa) or if the invasive reference diastolic range is more than 12 mmHg (1, 6 kPa) in any single determination.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2019-09-10 (Actual); Study Completion 2019-09-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Greta Piper, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: Data will be available upon reasonable request. Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Patients in SICU
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Patients in SICU
Number analyzed (Participants) | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.6 (16.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 0
  More than one race | 0
  Unknown or Not Reported | 4
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Average Error in Blood Pressure Readings
Description: If the value obtained from the LiveMetric determination lied within the range of the reference BP, an error of 0 mm Hg (0kPa) was assigned to this determination. If the value obtained from the LiveMetric determination lies outside the range of the reference BP, the value of the determination from the adjacent limit of the range of the variation of BP was subtracted. That difference represents the error for this determination.
  The arithmetic mean of the error is calculated and its experimental standard deviation from the errors of each recording for each BP value (Systolic & Diastolic) and determination for each patient.
Time Frame: during intervention for 30 minutes
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Patients in SICU
Number analyzed (Participants) | 8
mmHg
  Systolic | -1.5 (6.3)
  Diastolic | 3.2 (6.0)

ADVERSE EVENTS:
Time Frame: during intervention for 30 minutes
Arm/Group | Patients in SICU
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-18): https://cdn.clinicaltrials.gov/large-docs/35/NCT03629535/Prot_SAP_000.pdf